CLINICAL TRIAL: NCT02923440
Title: Creation of a French South-Eastern Database and DNA-bank of Congenital Heart Disease to Explore the Genetic Pathways
Acronym: SEA-HD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A00958-43; 2016-13 (Other: AP HM)
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Congenital Heart Defects
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Congenital heart defects (Experimental)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample

SUMMARY:
Congenital heart defects are seen in 0,8% of life births. In France this means more than 5000 newborns per year. The south-east region of France is particularly affected as a result of a higher birth rate and consanguinity, when compared to other regions. The majority of congenital heart diseases remain unexplained. Genetic causes are indisputable but remain poorly understood. Genetic research needs the availability of a large-scale DNA collection, guided by a robust phenotypic classification. Such a DNA-bank has been created in Paris (CARREG DNA bank, created by the M3C reference centre for congenital heart diseases). Such a bank is currently unavailable in south-east France. To transport biological specimens from Marseille to Paris would be very expensive. In addition, the whole infrastructure required for correct diagnosis and classification of the congenital heart diseases, for sampling, for storage of the samples and genetic analysis, does exist in our AP-HM hospital and in our AMU research unit. For those reasons it is highly preferable to elaborate such a database and DNA-bank locally. The acronym SEA-HD (South-EAst-Heart-Diseases) would be used to name this DNA-bank

ELIGIBILITY:
Inclusion Criteria:

* Echocardiographic diagnosis of congenital heart defect falling within the classification Houyel and Bonnet
* Necessity of making a blood test regardless of study
* Medical care in the AP-HM Timone Hospital children, medical-surgical unit of pediatric and congenital cardiology, Marseille - These Parent Child

Exclusion Criteria:

* Pregnant women
* Patients or parent / legal guardian (if minor) in physical or mental incapacity to understand or sign the consent
* People in Emergencies
* Persons deprived of freedom
* Persons not beneficiaries of a social security scheme
* Persons in health or social institution

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-01-17 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
number of patient with Congenital Heart Defects | 3years

CONTACTS AND LOCATIONS:
Overall Officials: catherine GEINDRE, Study Director — ASSISTANCE PUBLIQUE HÔPITAUX DE MARSEILLE
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No